CLINICAL TRIAL: NCT04957498
Title: Feasibility of Conducting a Randomized Controlled Trial Comparing Standard FBT and Guided Self-Help FBT for Adolescent Anorexia Nervosa
Brief Title: Feasibility Study Comparing Standard FBT and Guided Self-Help FBT for Adolescent Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Child Psychiatry and Pediatrics in the Department of Psychiatry and Behavioral Sciences and Director of the Eating Disorder Program for Children and Adolescents, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43195
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Anorexia Nervosa
Keywords: FBT; Family Based Treatment; Guided Self-Help
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT (Active Comparator): Family Based Treatment (FBT) includes up to 15 session (50-60 minutes) with a trained therapist.
  Interventions: Behavioral: Family Based Treatment
- FBT-GSH (Experimental): Family Based Treatment Guided Self-Help (FBT-GSH) includes an online website with educational videos, readings, discussion groups, and journals. Parents assigned to this arm will have up to 12 coaching sessions (20-30 minutes) with a trained therapist.
  Interventions: Behavioral: Guided Self-Help for Family Based Treatment

INTERVENTIONS:
Behavioral: Guided Self-Help for Family Based Treatment — A online website provided to parents containing information learned in Family Based Treatment and up to 12 coaching sessions with a therapist.
  Other Names: FBT-GSH
  Arms: FBT-GSH
Behavioral: Family Based Treatment — Standard Family Based Treatment provided for up to 15 sessions.
  Other Names: FBT
  Arms: FBT

SUMMARY:
This study examines a parent only Guided Self-Help for Family Based Treatment (GSH-FBT) for adolescents between the ages of 12 and 18 diagnosed with Anorexia Nervosa. Preliminary data collected in a previous study suggest that a Guided Parental Self-Help Version of FBT (GSH-FBT) has similar outcomes as therapist provided FBT.

DETAILED DESCRIPTION:
In this study, families will be randomized to either receive 12 weekly online sessions of Guided Self-Help for Family Based Treatment (GSH-FBT), or 15 sessions of online, professionally delivered, standard FBT over the course of 6 months. Potential subjects will be recruited from Stanford University, McMaster University, other local medical programs and clinics, and online advertisement to the population at large. If participants are deemed eligible, participants will be invited for a baseline interview during which the investigators will conduct interviews and collect questionnaire measures. Participants will complete a follow-up interview at the end of treatment and 3-month after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are 12-18 years of age
2. Participants live with a family (some families may contain only one parent)
3. Family members fluently speak and read English and have access to a computer with internet
4. Participants meet DSM-5 criteria for AN (both subtypes)
5. IBW between 75% and 88%
6. Participants are medically stable for outpatient treatment according to the recommended thresholds of the American Academy of Pediatrics and the Society of Adolescent Medicine
7. Participants are not engaged in another individual or family based psychotherapy trial during the duration of treatment sessions in the study.
8. Medications for comorbid psychiatric disorders are OK; randomization will balance groups through tracking.

Exclusion Criteria:

1. Associated physical illness that necessitates hospitalization
2. Psychotic illness in any form, mental retardation, autism, or any other mental illness that would interfere with the use of psychotherapy.
3. Current dependence on drugs or alcohol
4. Physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
5. Previous (5 or more sessions of) or current FBT-AN
6. Participants and family members do not have an adequate understanding of spoken English and are not able to speak and read English in order to participate in family therapy and the assessments.
7. Current weight is less than 75% or above 88% of expected weight given age and height.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Stanford University, Stanford, California, United States
- McMaster University, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- FBT-V: Family Based Treatment (FBT) includes up to 15 session (50-60 minutes) with a trained therapist.
  Family Based Treatment: Standard Family Based Treatment provided for up to 15 sessions.
- GSH-FBT: Family Based Treatment Guided Self-Help (FBT-GSH) includes an online website with educational videos, readings, discussion groups, and journals. Parents assigned to this arm will have up to 12 coaching sessions (20-30 minutes) with a trained therapist.
  Guided Self-Help for Family Based Treatment: A online website provided to parents containing information learned in Family Based Treatment and up to 12 coaching sessions with a therapist.
Period: Overall Study
Arm/Group | FBT-V | GSH-FBT
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FBT-V | GSH-FBT | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.93 (1.82) | 14.82 (1.86) | 14.88 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 18 | 35
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9 | 10 | 19
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Number of participants enrolled in the study per month.
Time Frame: Assessed through the end of recruitment (about one year)
Population: Since this is a feasibility study, all enrolled and randomized participants are analyzed together to report the rate that they were recruited to the study.
Measure: Number; unit: participants recruited per month
Groups:
- Overall Sample: Participants enrolled and randomized to a treatment arm (FBT-V or GSH-FBT).
Arm/Group | Overall Sample
Number analyzed (Participants) | 40
participants recruited per month | 2.86

2. Primary Outcome: Treatment Retention Rate
Description: The count of participants who did not stop treatment before finishing their randomized treatment course (FBT-V or GSH-FBT).
Time Frame: Up to 6 months
Population: Since this is a feasibility study, all participants who were enrolled and randomized to a treatment arm are analyzed together to report the treatment retention rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 40
Participants | 35

3. Primary Outcome: Study Retention Rate
Description: The number of participants who provided information for the end of treatment assessment and 3-month follow up assessment.
Time Frame: Up to 9 months
Population: Since this is a feasibility study, participants enrolled and randomized to a treatment arm are analyzed together to report the study retention rate.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Sample: Participants enrolled and randomized to a treatment arm.
Arm/Group | Overall Sample
Number analyzed (Participants) | 40
Participants | 37

4. Primary Outcome: Treatment Acceptability Ratings
Description: To assess treatment acceptability, the study used the Cooperation and Helpfulness sub-scales of the Helping Alliance Questionnaire (HAQ). The HAQ was administered to parents after session 1 and 8. The subscales, Helpfulness and Cooperation, are scored on a Likert scale from "Strongly feels it's true" (+3) to "Strongly feel it's not true" (-3). The sub-scales' total scores ranges are 15- to 15 for Helpfulness and -18 to 18 for Cooperation. A higher score indicates a better outcome. The average score was calculated if more than one parent responded.
Time Frame: Session 1 and Session 8 (approximately 5 minutes to complete questionnaire)
Population: Intent-to-treat population (excluding participants who were withdrawn from the study per investigator decision).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FBT-V | GSH-FBT
Number analyzed (Participants) | 20 | 18
score on a scale
  HAQ - Helpfulness after Session 1 | 3.97 (3.64) | 4.78 (4.75)
  HAQ - Helpfulness after Session 8 | 6.01 (4.36) | 7.77 (4.40)
  HAQ - Cooperation after Session 1 | 11.47 (3.30) | 11.91 (5.74)
  HAQ - Cooperation after Session 8 | 13.09 (3.68) | 12.38 (4.80)

5. Primary Outcome: Treatment Acceptability Ratings
Description: To assess treatment acceptability, the study used the Therapist Suitability and Patient Expectancy measure (TSPE). The TSPE was administered to parents after session 1. The scale is measured from 0-10 (with 0 as the lowest rating and 10 as the highest rating). The average score was calculated if more than one parent responded. A higher score on the TSPE indicates a better outcome.
Time Frame: Session 1 (approximately 5 minutes to complete questionnaire)
Population: Intent-to-treat population (excluding participants who were withdrawn from the study per investigator decision).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FBT-V | GSH-FBT
Number analyzed (Participants) | 20 | 18
score on a scale
  TSPE - Suitability of Treatment after Session 1 | 8.5 (1.37) | 7.85 (1.98)
  TSPE - Expectations of Therapy after Session 1 | 8.29 (1.29) | 7.35 (1.77)

6. Primary Outcome: Number of Treatment Sessions Attended
Description: The number of sessions completed by the the participant with the client in treatment is the actual, not planned, number of sessions actually conducted.
Time Frame: Through end of treatment (up to approximately 6 months)
Population: Intent-to-treat population (excluding participants who were withdrawn from the study per investigator decision).
Measure: Mean (Standard Deviation); unit: Sessions attended per participant
Arm/Group | FBT-V | GSH-FBT
Number analyzed (Participants) | 20 | 18
Sessions attended per participant | 13.32 (3.32) | 11.71 (0.77)

7. Primary Outcome: Serious Adverse Events
Description: Number of events in which a participant required hospitalization
Time Frame: Baseline through end of treatment period (up to 6 months)
Population: Following intent-to-treat principles, the number analyzed is based on the total N per sample in each arm, except for investigator withdrawals.
Measure: Number; unit: events
Arm/Group | FBT-V | GSH-FBT
Number analyzed (Participants) | 20 | 18
events | 2 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 9 months
Arm/Group | FBT-V | GSH-FBT
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 4/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FBT-V (N=20) | GSH-FBT (N=20)
Hospitalization (Psychiatric disorders) | 1 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04957498/Prot_SAP_000.pdf